CLINICAL TRIAL: NCT05270135
Title: ASAP: Access to Syringes at Pharmacies for the Prevention of Bloodborne Infections Among People Who Inject Drugs
Acronym: ASAP
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Arizona (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: 2011214920
Record Dates: First submitted 2022-02-15; First posted 2022-03-08 (Actual); Last update posted 2023-12-19 (Actual); Status verified 2023-12

CONDITIONS: Skin and Soft Tissue Infections; Hiv; Hepatitis C; Bloodstream Infection
MeSH Terms: conditions — Soft Tissue Infections; Acquired Immunodeficiency Syndrome; Hepatitis C; Sepsis

STUDY DESIGN:
Intervention Model Description: Pilot study of an intervention using one group comprised of three pharmacies and their enrolled staff.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- ASAP Intervention (Other): This is a pilot study of the ASAP intervention pharmacies to explore the preliminary impact of intervention components: the CEU training, coaching from research staff, ASAP materials and tracking for the sale of syringes. Staff of each enrolled pharmacy will complete surveys.
  Interventions: Behavioral: ASAP

INTERVENTIONS:
Behavioral: ASAP — ASAP is an intervention geared toward increasing non-stigmatized syringe sales to people who inject drugs to prevent bloodborne illnesses.

SUMMARY:
Access to Syringes at Pharmacies (ASAP) is a refinement of an evidence-based, pharmacy intervention to increase pharmacy-based sales of syringes to PWID in order to reduce bloodborne illnesses among them.

DETAILED DESCRIPTION:
The refinement integrates a motivational enhancement to reduce staff ambivalence about syringe sales to PWID (People who inject drugs), sampling improvements to assure that project pharmacies are likely serving PWID, and refinements to the intervention training content and delivery in three selected Arizona project counties of Mohave, Maricopa and Pima. Our development and refinement of ASAP relies on: 1) interviews with pharmacy staff of 6 pharmacies (2 for each county) that will assess feasibility, acceptance and likely adoption of the initial draft of the ASAP intervention, and 2) interviews and surveys among pharmacy staff of 3 pharmacies (1 from each county). ASAP's adaptations and refinements will be guided by a highly iterative process between investigators and a community advisory board (CAB). Further, the Consolidated Framework for Implementation Research (CFIR) will guide feasibility assessment with a focus on selected CFIR elements across the domains of intervention characteristics, outer and inner setting, characteristics of individuals and process. The project will occur in two phases. The Year 1 formative phase and is NOT a clinical trial will involve: 1) in-depth interviews with staff of 6 pharmacies to clarify intervention components, training and feasibility. Findings will inform the Year 2 iterative ASAP development and refinement phase and beta testing (clinical trial) between investigators and the CAB; including extensive feedback from pharmacy staff of 3 pharmacies following an ASAP beta test. Specific Aims are: Aim 1: To conduct the formative research among pharmacy staff required to develop and beta test the ASAP intervention materials (e.g., training manual, manual of operations, evaluation protocols).

Aim 2: To determine the feasibility of the ASAP intervention relative to impact on pharmacy syringe related sales and pharmacy interactions with PWID at time of syringe buy request.

ELIGIBILITY:
Inclusion Criteria:

* full time pharmacy staff member as a pharmacist or a pharmacy technician in an Arizona pharmacy within the three study counties (Pima, Maricopa, Mohave)

Exclusion Criteria:

* not a full time pharmacy staff member

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 18 (Actual)
Dates: Start 2022-12-01 (Actual); Primary Completion 2023-06-30 (Actual); Study Completion 2023-09-30 (Actual)

PRIMARY OUTCOMES:
Syringe sales increase as measured by the sales tracking instrument | by end of year 2
  ASAP pharmacies will increase the sale of nonprescription syringes upon request
Reduced stigma as measured by the feasibility assessment tool | by end of year 2
  ASAP pharmacy staff will report a reduction in expressed stigma at the time of syringe sales.

CONTACTS AND LOCATIONS:
Locations (1):
- University of Arizona College of Medicine, Tucson, Arizona, United States

IPD SHARING:
Plan to Share IPD: No